CLINICAL TRIAL: NCT03203057
Title: Serial Measurements of High-sensitivity Cardiac Troponin T and Troponin I After Short, Controlled Induced Cardiac Ischemia
Brief Title: Induced Myocardial Ischemia: a Serial Troponin T and Troponin I Measurements
Acronym: ICE-land
Status: Completed | Type: Observational
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Asthildur Arnadottir, Medical Doctor, Herlev Hospital
Other Study IDs: H-16027749
Record Dates: First submitted 2017-06-20; First posted 2017-06-29 (Actual); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Acute Coronary Syndrome; Cardiac Ischemia
MeSH Terms: conditions — Acute Coronary Syndrome; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- control group: 10 individuals get randomised to control group.
- short ischemic time: 10 individuals get randomised to a controlled coronary occlusion for 30 seconds
  Interventions: Other: coronary occlusion
- intermediate ischemic time: 10 individuals get randomised to a controlled coronary occlusion for 60 seconds
  Interventions: Other: coronary occlusion
- long ischemic time: 10 individuals get randomised to a controlled coronary occlusion for 90 seconds
  Interventions: Other: coronary occlusion

INTERVENTIONS:
Other: coronary occlusion — percutaneous coronary intervention
  Groups: intermediate ischemic time; long ischemic time; short ischemic time

SUMMARY:
Background Troponin are proteins found in the cardiomyocyte and are a cornerstone in the diagnoses of acute myocardial infarction. Troponin is released to the bloodstream as a result of an cardiomyocyte injury. Troponin is frequently assessed in hospital care for patients with chest pain and dyspnea.

Guidelines recommend troponin assessment at admission and repeated at 3 to 6 hours, depending on the assay. High-sensitivity assays measure concentrations that are ten-times lower than earlier generations of assays. However, the time from when troponin is elevated in the bloodstream after an ischemic injury, measured with high-sensitivity assays, are not fully known.

During an X-ray imaging of the heart's blood vessels (coronary angiogram) it is possible to do a short, controlled occlusion of coronary artery by inflating a small balloon in one of the coronary arteries. Numerous earlier studies in patients have used this method for induced occlusion of one coronary artery for 1 to 3 minutes. Only one of the studies measured troponin I.

The aim with this study is to quantify and compare the release of troponin T and troponin I in the early hours after a controlled induced ischemia.

Study Design This is a prospective, descriptive and experimental study. There will be included 40 patients, without acute ischemic cardiac disease. They will be randomized in 4 groups.

0: 10 patients - control group, no balloon occlusion

1. 10 patients - balloon occlusion for 30 seconds
2. 10 patients - balloon occlusion for 60 seconds
3. 10 patients - balloon occlusion for 90 seconds

Subsequently there will be assessed serial blood samples 0 - 3 hours: Every 15 minutes 3 - 6 hours: Every 30 minutes

Statistics This is a pilot study and it is estimated that ten patients are sufficient number of patients in each group to assess elevation of troponin after occlusion of coronary artery. The thesis is there is a dosage-response correlation between the length of balloon occlusion and the concentration of troponin in blood stream.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age Elective coronary angiogram Informed signed accept

Exclusion Criteria:

* Stenosis or atherosclerosis of the coronary artery Renal Failure or p-creatinin > 100 µmol/L Heart Failure or LVEF < 50 Severe Heart Valve Disease

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient referred to coronary angiography due to suspicion of ischemic heart disease.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2016-10-05 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
Troponin release | 6 hours
  Quantifying troponin T and I release after ischemic event

CONTACTS AND LOCATIONS:
Locations (1):
- Herlev-Gentofte Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arnadottir A, Pedersen S, Bo Hasselbalch R, Goetze JP, Friis-Hansen LJ, Bloch-Munster AM, Skov Jensen J, Bundgaard H, Iversen K. Temporal Release of High-Sensitivity Cardiac Troponin T and I and Copeptin After Brief Induced Coronary Artery Balloon Occlusion in Humans. Circulation. 2021 Mar 16;143(11):1095-1104. doi: 10.1161/CIRCULATIONAHA.120.046574. Epub 2020 Dec 10. PMID 33297742